CLINICAL TRIAL: NCT00632047
Title: Early Detection of Common Cancers in Women in India
Brief Title: Early Detection of Breast Cancer and Cervical Cancer in Women in India
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Screening
Other Study IDs: CDR0000586791; TATA-1900215717A1
Record Dates: First submitted 2008-03-07; First posted 2008-03-10 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer; Cervical Cancer
Keywords: breast cancer; cervical cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms | interventions — Watchful Waiting; Early Intervention, Educational; Restraint, Physical

INTERVENTIONS:
Other: active surveillance
Other: educational intervention
Procedure: examination
Procedure: long-term screening

SUMMARY:
RATIONALE: Health education programs and screening methods, such as clinical breast examination and examination of the cervix, may help reduce the number of women who develop breast cancer and cervical cancer.

PURPOSE: This randomized clinical trial is studying the early detection of breast cancer and cervical cancer in women in India.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the effectiveness of well planned health education programs (HEP) and low-cost screening methods (e.g., clinical breast examination [CBE] and visual inspection of the cervix painted with 4% acetic acid [VIA]) in down-staging and reducing the incidence of and mortality due to breast and cervical cancer.

OUTLINE: Patients are randomized to 1 of 2 arms.

* Arm I (intervention): Participants undergo intervention comprising health education programs (HEP), clinical breast examination (CBE), and visual inspection of the cervix painted with 4% acetic acid (VIA) every 2 years for up to 8 years. Participants also undergo active surveillance over 8 years.
* Arm II (control): Participants receive one HEP. Participants also undergo active surveillance over 8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Resides in 1 of 20 geographically defined clusters within the slums of Mumbai, India

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151538 (Estimated)
Dates: Start 1998-05; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of well planned health education programs and low-cost screening methods (e.g., clinical breast exam and visual inspection of the cervix) in reducing the incidence of and mortality due to breast and cervical cancer

CONTACTS AND LOCATIONS:
Overall Officials: Surendra S. Shastri, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, India

REFERENCES:
- [Result] Dinshaw K, Mishra G, Shastri S, Badwe R, Kerkar R, Ramani S, Thakur M, Uplap P, Kakade A, Gupta S, Ganesh B. Determinants of compliance in a cluster randomised controlled trial on screening of breast and cervix cancer in Mumbai, India. 1. Compliance to screening. Oncology. 2007;73(3-4):145-53. doi: 10.1159/000126497. Epub 2008 Apr 11. PMID 18408401
- [Result] Dinshaw K, Mishra G, Shastri S, Badwe R, Kerkar R, Ramani S, Thakur M, Uplap P, Kakade A, Gupta S, Ganesh B. Determinants of compliance in a cluster randomised controlled trial on screening of breast and cervix cancer in mumbai, India. 2. Compliance to referral and treatment. Oncology. 2007;73(3-4):154-61. doi: 10.1159/000126498. Epub 2008 Apr 11. PMID 18408402
- [Derived] Mittra I, Mishra GA, Dikshit RP, Gupta S, Kulkarni VY, Shaikh HKA, Shastri SS, Hawaldar R, Gupta S, Pramesh CS, Badwe RA. Effect of screening by clinical breast examination on breast cancer incidence and mortality after 20 years: prospective, cluster randomised controlled trial in Mumbai. BMJ. 2021 Feb 24;372:n256. doi: 10.1136/bmj.n256. PMID 33627312